CLINICAL TRIAL: NCT07374666
Title: The Effectiveness of a Mindfulness Based Program on Short- Form Video Addiction in Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Buse SAYGIN ŞAHİN, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/306
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Adolescence; Mindfulness; Addiction; Mental Health
Keywords: adolescence; mindfulness; addiction; mental health
MeSH Terms: conditions — Behavior, Addictive; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study is planned to include randomized intervention and control groups, with pre-test, post-test, and a follow-up assessment conducted three months after the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The study will be conducted with high school students. Those who provide informed assent, along with parental informed consent, will complete pre-test questionnaires. Students scoring above the average on the Short Video Addiction Scale will be randomly assigned to either the intervention group or the control group. The intervention group will participate in an 8-week mindfulness-based program, consisting of one session per week. A post-test will be administered at the end of the 8-week program, and follow-up assessments will be conducted three months after the intervention is completed.
  Interventions: Behavioral: Mindfulness Based Program
- Control Group (No Intervention): Students who provide informed assent, along with parental informed consent, will complete pre-test questionnaires. Those who score above the average on the Short Video Addiction Scale will be randomly assigned to either the intervention group or the control group. No intervention will be applied to the control group. Follow-up assessments will be conducted at the end of the 8-week period and again three months later.

INTERVENTIONS:
Behavioral: Mindfulness Based Program — The program will last for 8 weeks, with one session held each week. Each session will focus on specific themes such as mindfulness, acceptance, and compassion. The sessions include explanations of these concepts as well as practical exercises like breath awareness and body scan. At the end of each week, participants will be assigned homework to help reinforce their practice.
  Session Outline:
  Session 1: Introduction and Mindfulness
  Session 2: Sensations
  Session 3: The Wandering Mind
  Session 4: Challenges in Daily Life
  Session 5: Reactions
  Session 6: Compassion
  Session 7: Acceptance
  Session 8: Sustainability and Maintaining Practice
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a mindfulness-based program in reducing short form video addiction among adolescents. The study is designed as a randomized controlled trial with a pre-test, post-test, and follow-up design, including an intervention group and a control group.

Research Hypothesis:

Adolescents who participate in the Mindfulness-Based Program will have significantly lower short video addiction scores compared to those in the control group.

DETAILED DESCRIPTION:
In recent years, the widespread use of social media platforms that allow users to create and consume short videos has raised concerns regarding their addictive potential. The rapid, attention-grabbing, and entertaining nature of short video content is believed to intensify reinforcement mechanisms that lead to excessive screen time and addictive behaviors. These platforms offer instant gratification, enhance the flow experience, and contribute to behavioral patterns such as "phubbing"-the act of ignoring one's surroundings and social interactions in favor of smartphone use.

Among adolescents, this trend is particularly alarming. Adolescents constitute the largest user group of short video platforms and are more susceptible to the negative impacts of such content. Excessive short video use has been associated with various adverse outcomes, including decreased academic performance, impaired sleep quality, reduced physical health, poor self-control, and the development of psychological issues. Additionally, perceived stress has been identified as a significant risk factor contributing to short video addiction, especially among students.

Mindfulness, defined as the ability to maintain a moment-to-moment awareness of one's experiences with an open and non-judgmental attitude, has emerged as a promising approach in addressing behavioral addictions. Mindfulness-based practices are known to improve emotional regulation, reduce stress and anxiety, enhance self-awareness, and support academic performance. As such, mindfulness has been proposed as a protective factor against internet and technology-related addictions.

This study aims to examine the effectiveness of a mindfulness-based intervention in reducing short form video addiction among adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Being a 10th-grade high school student
* Having no visual, auditory, or comprehension impairments.
* Scoring above the mean on the Short Video Addiction Scale.
* Not being in a period close to exam time

Exclusion Criteria:

* Failure to attend two consecutive sessions
* Incomplete completion of research-related forms.
* Withdrawal from the study at any stage.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Short Video Addiction Scale | Pre-test, Post-test (8th week), Follow-up Test (12th week)
  The Short Video Addiction Scale, developed by Ye et al. (2022), aims to identify addiction, negative emotions, and experiences associated with watching short videos. The scale is unidimensional, consists of ten items, and uses a five-point Likert-type format. There are no reverse-scored items. Higher total scores indicate higher levels of addiction. The Turkish validity and reliability study of the scale was conducted by Türk and Yıldırım (2024), and the internal consistency coefficient of the scale was reported as 0.82.

SECONDARY OUTCOMES:
Short Video Flow Scale | Pre-test, Post-test (8th week), Follow-up Test (12th week)
  The Short Video Flow Scale was developed by Ye et al. and consists of eight items under a single dimension. This five-point Likert-type scale is designed to assess experiences such as watching and enjoying short videos. No items are reverse-scored. Higher total scores indicate greater enjoyment and longer viewing durations of short videos. Sample items include: "I can get lost while watching short videos and continue watching without realizing how time passes" and "I get so absorbed in the videos that I lose track of time." The Turkish validity and reliability study of the scale was conducted by Türk and Yıldırım (2024), and its internal consistency coefficient was 0.87.
General Phubbing Scale - Short Form | Pre-test, Post-test (8th week), Follow-up Test (12th week)
  the General Phubbing Scale - Short Form, developed by Li (2022) to evaluate phubbing behavior, was chosen for use in the present study. The Turkish validity and reliability study for adolescents was conducted by Kaya et al. (2024). The scale consists of 12 items under four subdimensions-nomophobia (e.g., "I can't stand being away from my phone"), interpersonal conflict (e.g., "I get annoyed when others ask me to put down my phone and talk to them"), self-isolation (e.g., "I feel good when I stop focusing on others and engage with my phone"), and problem acknowledgment (e.g., "When I use my phone, I often find myself thinking 'just a few more minutes'"). It is a seven-point Likert-type scale, with total scores ranging from 12 to 84; higher scores indicate higher levels of phubbing behavior. Reliability evidence was supported by Cronbach's alpha and McDonald's omega coefficients, while model fit indices were reported as RMSEA = .051-.084, CFI = .933-.975, NNFI/TLI = .912-.968.

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Sukut, PhD, Study Director — Istanbul University - Cerrahpasa
Locations (2):
- Turkey (Türkiye) (2):
  - High School - Site 1, Istanbul
  - High School - Site 2, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu, C., Jiang, Y., Lei, H., Wang, H., Zhang, C. 2024. "The relationship between short-form video use and depression among Chinese adolescents: Examining the mediating roles of need gratification and short-form video addiction", Heliyon, 10(9).
- [Background] Zhang, Y., Bu, R., Zhao, J., Li, X. 2023. "Social exclusion and short video addiction in Chinese college students: the mediating role of boredom and self-control", https://doi.org/10.21203/rs.3.rs-3654644/v1
- [Background] Xie, J., Xu, X., Zhang, Y., Tan, Y., Wu, D., Shi, M., Huang, H. 2023. "The effect of short-form video addiction on undergraduates' academic procrastination: a moderated mediation model", Frontiers in Psychology, 14, 1298361.
- [Background] Wu, A. 2023. "Communication psychology and short video communication on urban culture and social anxiety disorder in Chongqing", CNS Spectrums, 29-30.
- [Background] Wang, X., Zhao, S., Zhang, M. X., Chen, F., Chang, L. 2021. "Life history strategies and problematic use of short-form video applications", Evolutionary Psychological Science, 7, 39-44.
- [Background] Wang, H., Lei, L. 2022. "The relationship between parental phubbing and short-form videos addiction among Chinese adolescents", Journal of Research on Adolescence, 32(4), 1580-1591.
- [Background] Türk, N., Yıldırım, O. 2023. "Psychometric Properties of Turkish Versions of the Short Video Flow Scale and Short Video Addiction Scale", Bağımlılık Dergisi, 25(4), 384-397.
- [Background] Tian, X., Bi, X., Chen, H. 2023. "How short-form video features influence addiction behavior? Empirical research from the opponent process theory perspective", Information Technology & People, 36(1), 387-408.
- [Background] Sharma, M. K., Bhargav, H., Kumar, A., Digambhar, V., Mani, T. A. 2021. "Mindfulness-based interventions: potentials for management of internet gaming disorder", International Journal of Yoga, 14(3), 244-247.
- [Background] Shahmohammadi, N. 2011. "Students' coping with stress at high school level particularly at 11th & 12th grade", Procedia - Social and Behavioral Sciences, 30, 395-401.
- [Background] Pierce, B., Bowden, B., McCullagh, M., Diehl, A., Chissell, Z., Rodriguez, R., Berman, B. M. 2017. "A summer health program for African-American high school students in Baltimore, Maryland: community partnership for integrative health", Explore, 13(3), 186-197.
- [Background] Pharris-Ciurej, N., Hirschman, C., Willhoft, J. 2012. "The 9th grade shock and the high school dropout crisis", Social Science Research, 41(3), 709-730.
- [Background] Peng, C., Lee, J. Y., Liu, S. 2022. "Psychological phenomenon analysis of short video users' anxiety, addiction and subjective well-being", International Journal of Contents, 18(1), 27-39.
- [Background] Nong, W., He, Z., Ye, J. H., Wu, Y. F., Wu, Y. T., Ye, J. N., Sun, Y. 2023. "The relationship between short video flow, addiction, serendipity, and achievement motivation among Chinese vocational school students: the post-epidemic era context", Healthcare, 11(4), 462.
- [Background] Liu, Y., Ni, X., Niu, G. 2021. "Perceived stress and short-form video application addiction: a moderated mediation model", Frontiers in Psychology, 12, 747656.
- [Background] Kendirkıran, G., Bilgin, H. 2024. "The effect of mindfulness intervention on high school students' eating habits and body image perceptions", Current Psychology, 43(37), 29707-29723.
- [Background] Kaya, A., Şata, M., Türk, N., Özok, H. I., Yıldırım, M. 2024. "Reliability and Validity of Short-Form Generic Scale of Being Phubbed and Phubbing Among Turkish Adolescents and Young Adults", Journal of Technology in Behavioral Science, 1-8.
- [Background] Jiang, L., Yoo, Y. 2024. "Adolescents' short-form video addiction and sleep quality: the mediating role of social anxiety", BMC Psychology, 12(1), 369.
- [Background] Arıcı Özcan, N., Işıldar, H. K. 2021. "The effects of the mindfulness program on 12th-grade high school students' perceived stress, mindfulness, and self-efficacy levels", MOJES: Malaysian Online Journal of Educational Sciences, 9(3), 12-24.